CLINICAL TRIAL: NCT01360502
Title: Safety of Capsule Endoscopy Using Human Body Communication in Patients With Cardiac Pacemakers and Implantable Cardiac Defibrillators
Brief Title: Safety of Capsule Endoscopy in Patients With Implantable Cardiac Devices
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Si Young Song, Yonsei University College of Medicine
Other Study IDs: 1-2009-0021
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2009-09

CONDITIONS: Gastrointestinal Disease; Anemia
Keywords: capsule endoscopy; cardiac pacemaker; implantable cardiac defibrillator
MeSH Terms: conditions — Gastrointestinal Diseases; Anemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective study designed to assess safety and potential influence of the MiroCam on cardiac pacemaker and implantable cardiac defibrillator.

DETAILED DESCRIPTION:
MiroCam (IntroMedic, Ltd, Seoul, Korea) is a small bowel capsule endoscope using human body communication for data transmission. There is a concern of potential interactions between cardiac devices and capsule endoscope. This clinical study was designed to evaluate the potential influence of the MiroCam on cardiac pacemaker and implantable cardiac defibrillator.

ELIGIBILITY:
Inclusion Criteria:

1. age 20 years or older
2. cardiac pacemaker or implantable cardiac defibrillator
3. gastrointestinal disease

Exclusion Criteria:

1. previous GI perforation or obstruction history
2. known or suspected GI stricture
3. marked GI dysmotility
4. uncompensated heart failure (EF ≤30% or Killip's classification class ≥ III)
5. pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with implantable cardiac devices
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Si Young Song, M.D., Ph.D., Study Chair — Yonsei University
Locations (1):
- Severance Hospital, Seoul, South Korea